CLINICAL TRIAL: NCT04098952
Title: Effects of Electric Massage on the Cervical Region Combined With Local Techniques on the Temporomandibular Joint Versus an Intervention Only With Local Techniques in Subjects Diagnosed With Temporomandibular Disorders
Brief Title: Effects of Electric Massage on the Cervical Region in Subjects Diagnosed With Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Espejo Antúnez PhD (Other)
Responsible Party: Sponsor-Investigator, Luis Espejo Antúnez PhD, Department of Medical Surgical Therapy., Universidad de Extremadura
Organization: Universidad de Extremadura (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LE0001
Record Dates: First submitted 2019-06-10; First posted 2019-09-23 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Temporomandibular Disorders
Keywords: temporomandibular disorders; electric massage; temporomandibular joint; local techniques
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Manual Therapy (Active Comparator): The treatment techniques used will be: ischemic compression in the trigger point of the masseter and soft-tissue release technique over the temporal region.
  Interventions: Other: Group 1: Manual Therapy
- Group 2: Interferential massage plus Manual Therapy (Experimental): In addition to the treatment techniques applied to the other group, an electric massage will be performed with interferential currents at the level of the cervical region.
  Interventions: Other: Group 2: Interferential massage plus Manual Therapy

INTERVENTIONS:
Other: Group 1: Manual Therapy — The treatment techniques used will be: ischemic compression in the trigger point of the masseter and soft-tissue release technique over the temporal region.
  Arms: Group 1: Manual Therapy
Other: Group 2: Interferential massage plus Manual Therapy — In addition to the treatment techniques applied to the other group, an electric massage will be performed with interferential currents at the level of the cervical region.
  Arms: Group 2: Interferential massage plus Manual Therapy

SUMMARY:
To know the short-term effects of electric massage applied on the cervical region combined with local techniques on the temporomandibular joint versus an intervention that applies only local techniques in subjects diagnosed with temporomandibular disorders.

DETAILED DESCRIPTION:
This study aims to know the short-term effects of electric massage applied to the cervical region combined with local techniques on the temporomandibular pain versus an intervention that applies only local techniques in subjects diagnosed with temporomandibular disorders. This is a prospective, controlled, single-blind clinical trial of 46 subjects randomly divided into two groups: Group 1 Manual Therapy=21; Group 2 Interferential massage plus Manual Therapy=25. Group 1 will receive manual therapy consisting of techniques of ischemic compression on masseter muscles and soft-tissue release technique over the temporal región. Group 2, in addition to the intervention in group 1, will receive electric massage with interferential currents at the cervical level.

Pain related measures (Visual Analogue Scale oral, Pressure Pain Threshold (PPT)), vertical mouth opening as primary outcome measures and cervical range of motion as secondary outcomes were assessed. The assessments were made before the intervention, immediately after and after 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the subject to participate in the study.
* A primary diagnosis of myofascial pain according to Axis I, category Ia and Ib (i.e. myofascial pain with or without limited opening) of the Research Diagnostic Criteria for TMD (RDC ⁄ TMD) (Schiffman E, Ohrbach R, Truelove E, et al. Diagnostic criteria for tempormandibular disorders (DC(TMD) for clinical and research applications: recommendations of the International RDC/TMD consortium network* and orofacial pain special interest group. J Oral facial pain headache. 2014;28(1):6-27").
* Bilateral pain involving the masseter and temporal regions; presence of at least one trigger point (TrP) in the masseter muscle.
* Pain symptoms history of at least the 3 months previous to the study.
* Intensity of the pain of at least 30 mm on a 100 mm Visual Analogue Scale (VAS).
* A score of less than 45 points on the Personal Psychological Apprehension Scale (PPAS). It has been validated in the scope of physiotherapy, and represents a simple-to-handle tool in studies where subjects may undergo electrotherapy as a treatment option.

Exclusion Criteria:

* Surgical intervention of the temporomandibular joints (TMJ).
* Suffering some intra-articular damage (arthritis) or some vestibular disorder diagnosed.
* Inflammation of the TMJ.
* Having received physiotherapy treatment in the last two weeks.
* Receive pharmacological treatment for analgesic, anti-inflammatory or that could cause alterations of equilibrium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Changes in the assessment of the maximum amplitude of the vertical opening of the mouth: | Immediately after the intervention as well as 4 weeks after the intervention.
  The maximum vertical opening of the mouth was measured using a manual gauge. The measurements were taken with the subjects placed in the supine position on the stretcher, with the head resting on it, the cervical spine in a neutral position, knees slightly bent and the upper limbs extended along the body.
  In this position, we ask participants to open their mouths as much as possible without causing pain. In this way, we obtain the measurement in millimeters the distance between the upper and lower central incisors.
Changes in the assessment of pain intensity: VAS | Immediately after the intervention as well as 4 weeks after the intervention.
  To measure pain, the visual analog scale (VAS) has been used. The VAS scale is an instrument used very often to quantify the intensity of pain. The accuracy and validity of the EVA scale as a measure of pain has been demonstrated previously.
  Participants were asked to indicate the degree of pain intensity in response to manual palpation of the central trigger point of the masseter bilaterally using a 10 cm analogue visual scale where 0 corresponds to "no pain" and 10 to "worst pain" that you can imagine. " When performing the post-treatment assessment, a period of 1 minute of rest was left to prevent the change of position from influencing the data obtained, especially in the displacements of the pressure center.
Changes in the valuation of pain threshold to pressure. | Immediately after the intervention as well as 4 weeks after the intervention.
  To measure the pain threshold to the pressure in muscle trigger points, a manual algometer with 1 cm2 of contact area was used. The algometer serves to record the minimum amount of pressure needed for the sensation of pressure to change to a sensation of pain. When this moment arrives, the subject will say "already" and the algometer immediately withdrawn, the pressure being recorded. The results obtained will be expressed in kg / cm2 (1,8).
  The muscles assessed were masseter and superior trapezius, both bilaterally in the supine position. The pressure in both must be done in a direction perpendicular to the muscle fibers. In the case of the upper trapezius, the algometer will be placed on the trigger point 1 described by Travell and Simons (9). In the masseter, the pressure perpendicular to the algometer will be applied on the central trigger point of the superficial portion of said muscle as described by Travell.

SECONDARY OUTCOMES:
Changes in the assessment of cervical range of motion. | Immediately after the intervention as well as 4 weeks after the intervention.
  The goniometry is used to evaluate the range of joint movement. The range of cervical movement can be evaluated with many instruments, but the goniometer offers a simple and low cost alternative for evaluation.
  In this case, for the measurement of the range of cervical movement we will use a universal goniometer that presents a scale of measurement in degrees. The patient will be placed in a sitting position in a chair and we will give him the order to perform the movement to be evaluated. The movements to be evaluated will be right and left rotation, flexion, extension and right and left side bending. We will prevent the patient from making compensations with other body regions.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo Antúnez, PhD, Study Director — Department of Medical Surgical Therapy.
Locations (1):
- Luis Espejo Antúnez, Badajoz, Spain

REFERENCES:
- [Derived] Espejo-Antunez L, Cardero-Duran MLA, Heredia-Rizo AM, Casuso-Holgado MJ, Albornoz-Cabello M. Effects of adding electro-massage to manual therapy for the treatment of individuals with myofascial temporomandibular pain: a randomized controlled trial. J Appl Oral Sci. 2024 Sep 16;32:e20240109. doi: 10.1590/1678-7757-2024-0109. eCollection 2024. PMID 39292112